CLINICAL TRIAL: NCT05821530
Title: A Randomized Controlled Clinical Trial Evaluating the Effectiveness of High-frequency Impulse Therapy (HFIT) Versus Transcutaneous Electronic Nerve Stimulator (TENS) for Treatment of Chronic Low Back and Knee Pain
Brief Title: HFIT Versus TENS Study for Chronic Low Back and Knee Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hinge Health, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HFIT20223468
Record Dates: First submitted 2023-04-06; First posted 2023-04-20 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Chronic Pain; Knee Pain Chronic; Back Pain, Low
Keywords: musculoskeletal; chronic; pain; knee pain; back pain
MeSH Terms: conditions — Chronic Pain; Low Back Pain; Bronchiolitis Obliterans Syndrome; Pain; Back Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- HFIT (Experimental): Participants received a HFIT device to treat their chronic pain and took part in a digital MSK program, which provided customized exercise therapy sessions, educational articles, and access to coaches and physical therapists. Participants were encouraged to use the HFIT device for at least 1 hour daily for 4 weeks.
  Interventions: Device: HFIT
- TENS (Experimental): Participants received a TENS device to treat their chronic pain and took part in a digital MSK program, which provided customized exercise therapy sessions, educational articles, and access to coaches and physical therapists. Participants were encouraged to use the TENS device for at least 1 hour daily for 4 weeks.
  Interventions: Device: TENS
- Control (Active Comparator): Participants took part in a digital MSK program, which provided customized exercise therapy sessions, educational articles, and access to coaches and physical therapists.
  Interventions: Other: Control

INTERVENTIONS:
Device: HFIT — At least 1 hour daily for 4 weeks
  Other Names: Enso
  Arms: HFIT
Device: TENS — At least 1 hour daily for 4 weeks
  Arms: TENS
Other: Control — Users will continue to use the digital MSK program as needed
  Other Names: Digital MSK program
  Arms: Control

SUMMARY:
A high-frequency impulse therapy (HFIT) device (Enso, San Francisco, CA) is a portable device for the treatment of musculoskeletal pain. This three-arm randomized controlled trial study compares a HFIT group to a standard transcutaneous electrical nerve stimulator (TENS) group and a control group.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over and under age 65
* Baseline pain is 40 or more out of 100 on a NPRS
* Member of digital MSK program's chronic back or knee pain program, after January 1, 2023
* Member engaged in the most recent 3 weeks
* Experiencing chronic pain for at least 3 months
* Subject able to understand and provide informed consent
* Has an email account

Exclusion Criteria:

* Diagnosis of cancer/malignant tumors in the last 5 years
* Back or knee surgery in the last 6 months
* Has a cardiac pacemaker, implanted defibrillator, spinal cord stimulator, pain pump, insulin pump, or any other implanted electronic device
* Patients with history of opioid, alcohol, or drug abuse in the last 1 year
* Cognitive, behavioral, neurologic, or psychiatric disorder (e.g., dementia, Parkinson's, schizophrenia, stroke) that may interfere with the study or prevent the subject from complying with the requirements of the protocol
* Pregnant or plan on becoming pregnant in the next year
* Have epilepsy
* Have cardiovascular disease
* Current pain (in the past 24 hours) is less than 40 out of 100 on a NPRS

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 325 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain MCID | Baseline and Week 4
  Pain will be measured by the Numeric Pain Rating Scale, ranging from 0 (no pain) to 100 (worst possible pain). The minimal clinically important difference (MCID) of pain will be achieved (0/1) if there is at least a 34% or 23 point improvement, as based on literature.

SECONDARY OUTCOMES:
Function MCID (Back) | Baseline and Week 4
  Back function will be measured by the Roland-Morris Disability Questionnaire 11-item (RMDQ-11, 0-100, higher indicates worse function) scores for back users. Function MCID will be achieved (0/1) if there is at least a 30% improvement in RMDQ-11, as based on literature.
Function MCID (Knee) | Baseline and Week 4
  Knee function will be measured by the Knee Injury and Osteoarthritis Outcome Score - Physical Short Form (KOOS-PS, 0-100, higher indicates worse function). Function MCID will be achieved (0/1) if there is at least an 8 point improvement in KOOS-PS, as based on literature.
Anxiety | Baseline and Week 4
  Anxiety will be assessed by the Generalized Anxiety Disorder 2-item (GAD-2, 0-6, higher is worse) scores. A score of 3 or higher is defined as screening in for having anxiety, based on literature. The percentage of users who screen in for anxiety in each group will be compared.
Depression | Baseline and Week 4
  Depression will be assessed by the Patient Health Questionnaire 2-item (PHQ-2, 0-6, higher is worse) scores. A score of 3 or higher is defined as screening in for having depression, based on literature. The percentage of users who screen in for depression in each group will be compared.
Opioid use | Baseline and Week 4
  Opioid use data will be collected through survey questions. The percentage of users who use opioids in each group during the study will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Hinge Health, Inc, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No